CLINICAL TRIAL: NCT04875988
Title: Point of Care UltraSound (POCUS) Use for Intravenous Catheter Placement During Pediatric Interfacility Transport
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 262598
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Intravenous Access
Keywords: pediatrics; interfacility transport; intravenous access; ultrasound; POCUS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- POCUS-assisted IV placement (Active Comparator): using ultrasound to help with placement
  Interventions: Procedure: Butterfly iQ+ Ultrasound
- Traditional IV placement (Active Comparator): Standard of care
  Interventions: Procedure: Traditional

INTERVENTIONS:
Procedure: Butterfly iQ+ Ultrasound — ultrasound will be used in the intervention group for IV access
  Arms: POCUS-assisted IV placement
Procedure: Traditional — ultrasound will not be used in the traditional IV placement group
  Arms: Traditional IV placement

SUMMARY:
This study will determine the efficacy of POCUS (Point of Care UltraSound) for intravenous (IV) access during pediatric interfacility transport. The Butterfly iQ+ (Lightning) device will be used. Children requiring IV access for transport will be randomized to POCUS-Assisted IV placement or traditional IV placement. We will examine and compare first attempt success rates with each method.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients requiring IV access prior to transport by the Angel One Transport Team back to Arkansas Children's Hospital
* Age group: 2 weeks - 18 years

Exclusion Criteria:

* Adequate IV Access
* NICU transports
* Patients not needing IV access

Ages: 2 Weeks to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
First Attempt IV success rates | 1 day of transfer

SECONDARY OUTCOMES:
Beside Times during transport | up to 24 hours
  as reported (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Stroud, MD, Principal Investigator — University of Arkansas

IPD SHARING:
Plan to Share IPD: No